CLINICAL TRIAL: NCT05634733
Title: Evaluation of Mitral Annulus Systolic Plane Excursion (MAPSE) in Emergency Department Patients With Sepsis
Brief Title: Change in MAPSE During Treatment of Sepsis
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Alexis Salerno, Assistant Professor of Emergency Medicine, University of Maryland, Baltimore
Other Study IDs: HP-00102983
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Sepsis
Keywords: POCUS; Emergency Department; echocardiography
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Sepsis: These are patients who present to the emergency department with sepsis. They will have a MAPSE at the time of enrollment and then after initial treatment.
  Interventions: Other: Treatment of Sepsis

INTERVENTIONS:
Other: Treatment of Sepsis — Patients will have standard care of sepsis

SUMMARY:
Patients with bloodstream infections (sepsis) have been found in prior studies to have infection-related heart dysfunction, even if they did not have preexisting heart problems. Factors related to the infection may cause the heart to not pump as well as it should, causing critical illness in the form of low blood pressure (shock) and heart failure. Ultrasound is frequently used in the emergency department to evaluate why a patient might have low blood pressure. Part of that evaluation may include obtaining ultrasound images and making measurements about how well or poorly the heart is pumping. The investigators will evaluate a certain measurement that relates to cardiac function, determine how it changes in patients before and after they are treated for septic shock. This will involve placing an ultrasound probe on the patient's chest, measuring the upward and downward movement of the mitral valve, the mitral annulus systolic plane excursion (MAPSE), and comparing the measurements before and after treatment is started. The investigators are attempting to determine if this measurement improves before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sepsis or Septic Shock

Exclusion Criteria:

* Age equal to or less than 17
* patient in the emergency department
* Unable to perform POCUS exam due to medical necessity
* Patients without sepsis
* unable to obtain consent or have a legal representative consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult emergency department patients who present with sepsis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in MAPSE measurement | 1 hour after treatment initiation
  Does the MAPSE change after treatment of MAPSE

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No